CLINICAL TRIAL: NCT03932500
Title: Outcomes of Traumatic Brain Injury and External Validation of CRASH Prognostic Model in a Tertiary Care Public University Hospital
Brief Title: Outcomes of Traumatic Brain Injury and External Validation of CRASH Prognostic Model
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Seth Gordhandas Sunderdas Medical College (Other)
Responsible Party: Principal Investigator, Monty Khajanchi, Assistant Professor, Department of General Surgery, Seth Gordhandas Sunderdas Medical College
Other Study IDs: EC/198/2017; U1111-1231-3772 (Other: Universal Trial Registration)
Record Dates: First submitted 2019-04-25; First posted 2019-04-30 (Actual); Last update posted 2019-04-30 (Actual); Status verified 2019-04

CONDITIONS: Brain Injuries, Traumatic
Keywords: Validation; Prognostic score
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
As per World Health Organization (WHO) 2015 report, road injury is the tenth cause of mortality in the world.

* 90% of these occur in Low and Middle-Income countries (LMICs)
* Amongst Injuries, Traumatic Brain Injuries is the leading cause of morbidity and mortality.
* Clinicians have to answer about the prognosis of the injured patient to the anxious near ones on arrival as well as throughout the course of treatment
* A multicenter randomized control trial (CRASH)published a prediction model for traumatic brain injury patients
* This model was based on data from High Income countries and not from Low and Middle-Income Countries
* Hence to fill this gap we aim to study the outcome of patients with Traumatic Brain Injury and also validate the CRASH trial prediction model in traumatic brain injury patient
* It is a Prospective Observational Study for a duration of 18 months and the sample size is 500 patients.
* Acute Traumatic Brain injury patients >18 years of age admitted in Emergency surgery room.
* Patients with chronic head injury and Patients who have been declared brain dead and whose organs have been retrieved are excluded.
* Variable are Age, Glasgow coma score, Pupils reaction to light, Major extra cranial injuries, CT Finding.
* Outcome of the study is mortality at 14th day and morbidity and mortality after 6 months of head injury.

DETAILED DESCRIPTION:
Introduction As per World Health Organization (WHO) 2015 report, road injury is the tenth cause of mortality in the world[1]. 90% of these occur in Low and Middle-Income countries (LMICs)[2]. The complex interaction of human, vehicle and environmental factors along with lack of sustainable preventive programs has contributed to this 'silent epidemic' of injuries. Amongst Injuries, Traumatic Brain Injuries is the leading cause of morbidity and mortality.

The young working men of age 20-40 years are the most vulnerable group to suffer a Traumatic Brain Injury[3]. Around 60% of those with TBI do not resume work[3]. A study done in Delhi, India showed that patients with severe TBI who were unconscious at discharge, 50% of them died at six months and another 30% remained in vegetative state[4].

Clinicians have to answer about the prognosis of the injured patient to the anxious near ones on arrival as well as throughout the course of treatment. Researches have shown prognostic models are statistical models that combine data from patients to predict outcome are likely to be more accurate than simple clinical predictions[5]. A multicenter randomized control trial published a prediction model for traumatic brain injury patients[6]. Unlike other prediction models this model was based on data from High Income and Low Middle-Income Countries. However, the external validation of this prediction model was not done in LMICs data[7]. Hence to fill this gap we aim to study the outcome of patients with Traumatic Brain Injury and also validate the CRASH trial prediction model in traumatic brain injury patient. e.g. A 45 year old male , came with road traffic accident leading to traumatic brain injury. His Glasgow Coma Scale was E4V4M5, both the pupils reacting to light and CT scan brain suggestive of Sub-dural hematoma of thickness approximately 3 mm along left basi-frontal superior and middle frontal convexities without significant underlying mass effect. These details inserted in CRASH PROGNOSTIC MODEL calculator as shown below. As per this the mortality at 14 day is 4.4% and morbidity at 6th month is 12.6% i.e. unfavorable outcome.

Data collection Data collection will be done by a resident and a medical student of the same hospital. Patients will be prospectively followed in the ward till discharge or death. Information will be entered in the case record form based on patients file. Written, valid informed consent will be taken to follow up patients on day 14th day and 6 months after the date of injury by telephonic conversation.

Outcomes:

Outcome of the study is mortality at 14th day and mortality and morbidity at 6th months after head injury. This morbidity at 6th months will be measured by using GLASGOW OUTCOME SCALE by telephonic conversation

Variables:

Demographic Variables, mechanism of injury, transfer status, vital parameters on admission like systolic blood pressure, heart rate, Glasgow coma scale will be noted from case records. Patients pupillary response will be collected from case record sheet. Ct scan findings and whether or not patient was operated (neurosurgery) will be noted. Other injuries will also be recorded.

Sample Size The sample size for an external validation study should have at least 100 patients with the outcome and 100 without the outcomes[8,]. The short-term outcome is mortality at 14 days. The mortality in all groups of TBI is 23%. So, to have 100 events we will need a sample size of minimum 500 patients. An interim analysis will be done at one year to see if the sample size is met and a further decision on the study duration will be made.

Analysis Data will be entered in Microsoft Excel 2016 and statistical analysis will be done using SPSS version 17. We will assess the performance of the models in our dataset in terms of discrimination and calibration. Discrimination describes how well a model distinguishes between patients with and without the outcome of interest. Calibration indicates how closely predicted outcomes match observed outcomes.

To assess discrimination, we will calculate the area under the receiver operating characteristic curve (AUC). An AUC of 1 implies perfect discrimination, whereas an AUC of 0.5 implies that a model's discrimination is no better than chance.

To assess calibration, we will plot observed versus predicted outcome. Ethics Informed consent will be taken by the co-investigator of this study from the patient/relative (legal representative), after patient is admitted in the ward. The informed consent will be to follow up the patient telephonically at 14 days and 6 months from the date of injury. During course in ward or at discharge if patient is conscious and is in a state to give consent, re-consent will be taken from patient himself. If the patient refuses to give consent then his/her data will not be recorded and no follow up will be done for the purpose of study.

ELIGIBILITY:
Inclusion Criteria:

* Adults with age more than 18 years presenting with acute Traumatic Brain Injury to the emergency surgical services of King Edward Memorial Hospital, Parel, Mumbai and get admitted will be enrolled in the study.

Exclusion Criteria:

* Patients with chronic head injury will be excluded. Patients who have been declared brain dead and whose organs have been retrieved will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with age more than 18 years presenting with acute Traumatic Brain Injury to the emergency surgical services of King Edward Memorial Hospital, Parel, Mumbai and get admitted will be enrolled in the study.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2018-03-22 (Actual); Primary Completion 2019-06-30 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Mortality | 14 days

SECONDARY OUTCOMES:
Morbidity | 6 months
  The Glasgow Outcome Scale (GOS) is a global scale for functional outcome that rates patient status into one of five categories: Dead (1), Vegetative State (2), Severe Disability(3), Moderate Disability (4) or Good Recovery (5). 1 is the worst and 5 is the best.
Mortality | 6 months
  The Glasgow Outcome Scale (GOS) is a global scale for functional outcome that rates patient status into one of five categories: Dead (1), Vegetative State (2), Severe Disability(3), Moderate Disability (4) or Good Recovery (5). 1 is the worst and 5 is the best.

CONTACTS AND LOCATIONS:
Locations (1):
- Seth GS Medical College and KEM Hospital, Mumbai, Maharashtra, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Haagsma JA, Graetz N, Bolliger I, Naghavi M, Higashi H, Mullany EC, Abera SF, Abraham JP, Adofo K, Alsharif U, Ameh EA, Ammar W, Antonio CA, Barrero LH, Bekele T, Bose D, Brazinova A, Catala-Lopez F, Dandona L, Dandona R, Dargan PI, De Leo D, Degenhardt L, Derrett S, Dharmaratne SD, Driscoll TR, Duan L, Petrovich Ermakov S, Farzadfar F, Feigin VL, Franklin RC, Gabbe B, Gosselin RA, Hafezi-Nejad N, Hamadeh RR, Hijar M, Hu G, Jayaraman SP, Jiang G, Khader YS, Khan EA, Krishnaswami S, Kulkarni C, Lecky FE, Leung R, Lunevicius R, Lyons RA, Majdan M, Mason-Jones AJ, Matzopoulos R, Meaney PA, Mekonnen W, Miller TR, Mock CN, Norman RE, Orozco R, Polinder S, Pourmalek F, Rahimi-Movaghar V, Refaat A, Rojas-Rueda D, Roy N, Schwebel DC, Shaheen A, Shahraz S, Skirbekk V, Soreide K, Soshnikov S, Stein DJ, Sykes BL, Tabb KM, Temesgen AM, Tenkorang EY, Theadom AM, Tran BX, Vasankari TJ, Vavilala MS, Vlassov VV, Woldeyohannes SM, Yip P, Yonemoto N, Younis MZ, Yu C, Murray CJ, Vos T. The global burden of injury: incidence, mortality, disability-adjusted life years and time trends from the Global Burden of Disease study 2013. Inj Prev. 2016 Feb;22(1):3-18. doi: 10.1136/injuryprev-2015-041616. Epub 2015 Dec 3. PMID 26635210
- [Background] Gururaj G. Epidemiology of traumatic brain injuries: Indian scenario. Neurol Res. 2002 Jan;24(1):24-8. doi: 10.1179/016164102101199503. PMID 11783750
- [Background] Agrawal D, Singh PK, Sinha S, Gupta DK, Satyarthee GD, Misra MC. Remaining unconscious: The burden of traumatic brain injuries in India. J Neurosci Rural Pract. 2015 Oct-Dec;6(4):520-2. doi: 10.4103/0976-3147.165394. PMID 26752896
- [Background] Lee KL, Pryor DB, Harrell FE Jr, Califf RM, Behar VS, Floyd WL, Morris JJ, Waugh RA, Whalen RE, Rosati RA. Predicting outcome in coronary disease. Statistical models versus expert clinicians. Am J Med. 1986 Apr;80(4):553-60. doi: 10.1016/0002-9343(86)90807-7. PMID 3963036
- [Background] MRC CRASH Trial Collaborators; Perel P, Arango M, Clayton T, Edwards P, Komolafe E, Poccock S, Roberts I, Shakur H, Steyerberg E, Yutthakasemsunt S. Predicting outcome after traumatic brain injury: practical prognostic models based on large cohort of international patients. BMJ. 2008 Feb 23;336(7641):425-9. doi: 10.1136/bmj.39461.643438.25. Epub 2008 Feb 12. PMID 18270239
- [Background] Roozenbeek B, Lingsma HF, Lecky FE, Lu J, Weir J, Butcher I, McHugh GS, Murray GD, Perel P, Maas AI, Steyerberg EW; International Mission on Prognosis Analysis of Clinical Trials in Traumatic Brain Injury (IMPACT) Study Group; Corticosteroid Randomisation After Significant Head Injury (CRASH) Trial Collaborators; Trauma Audit and Research Network (TARN). Prediction of outcome after moderate and severe traumatic brain injury: external validation of the International Mission on Prognosis and Analysis of Clinical Trials (IMPACT) and Corticoid Randomisation After Significant Head injury (CRASH) prognostic models. Crit Care Med. 2012 May;40(5):1609-17. doi: 10.1097/CCM.0b013e31824519ce. PMID 22511138
- [Background] Collins GS, Ogundimu EO, Altman DG. Sample size considerations for the external validation of a multivariable prognostic model: a resampling study. Stat Med. 2016 Jan 30;35(2):214-26. doi: 10.1002/sim.6787. Epub 2015 Nov 9. PMID 26553135